CLINICAL TRIAL: NCT05997862
Title: A Hip Flexion Feedback System for Exercise Monitoring in Individuals With Osteoarthritis and Obesity
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern Mississippi (Other)
Responsible Party: Principal Investigator, Nuno Oliveira, Assistant Professor, University of Southern Mississippi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-0210
Record Dates: First submitted 2023-05-01; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis, Knee; Obesity
Keywords: Exercise; Osteoarthritis; Obesity
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity; Motor Activity; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will do a 12-week high intensity exercise program. The subjects will exercise by increasing how much they lift their knees while walking on treadmill. The exercise will also involve controlling the impact of the feet on the treadmill. A TV placed in front of the treadmill shows how high individuals need to lift their knees. How much participants need to lift their knees is calculated based on real-time heart rate readings.
  Interventions: Device: HFFS
- Control (No Intervention): This group will do initially a 12-week period of no intervention. After these 12 weeks, participants will do a 12-week high intensity exercise program. The subjects will exercise by increasing how much they lift their knees while walking on treadmill. The exercise will also involve controlling the impact of the feet on the treadmill. A TV placed in front of the treadmill shows how high individuals need to lift their knees. How much participants need to lift their knees is calculated based on real-time heart rate readings.

INTERVENTIONS:
Device: HFFS — This study introduces a new way to exercise using a hip flexion feedback system (HFFS). The subjects will exercise by increasing how much they lift their knees while walking on treadmill. The exercise will also involve controlling the impact of the feet on the treadmill. The HFFS monitors the subject's heart rate during the exercise using a standard heart rate monitor. A TV placed in front of the treadmill shows how high individuals need to lift their knees. How much participants need to lift their knees is calculated by the HFFS based on real-time heart rate readings. Therefore, the HFFS can help people stay at a specific exercise intensity by controlling how high it tells them lift their knees during the exercise.
  Arms: Intervention

SUMMARY:
Exercise is very important for living healthier and longer lives. For people with obesity and osteoarthritis, exercise is even more important because it can help them feel less pain in their joints. Also, the more intense the exercise is, the larger the health benefits will be. The most common ways to exercise are running and riding a stationary bicycle. However, these two types of exercise can cause problems for people with obesity and osteoarthritis. Fast running creates large loads in the knees because of the impact of the foot on the ground. On the other hand, studies in cycling show limited improvement in pain because cycling does not allow the feet to move freely, which is important for reducing pain in people with osteoarthritis. This study introduces a new way to exercise using a hip flexion feedback system (HFFS). The subjects will exercise by increasing how much they lift their knees while walking on treadmill. The exercise will also involve controlling the impact of the feet on the treadmill. The HFFS monitors the subject's heart rate during the exercise using a standard heart rate monitor. A TV placed in front of the treadmill shows how high individuals need to lift their knees. How much participants need to lift their knees is calculated by the HFFS based on real-time heart rate readings. Therefore, the HFFS can help people stay at a specific exercise intensity by controlling how high it tells them lift their knees during the exercise. This study will have participants with osteoarthritis and obesity in two groups. One group will exercise using the HFFS. Another group will not exercise. The exercise group will do a 12-week high intensity exercise program. Our first goal is to determine how much fitness, pain, and the ability to move improve due to the exercise program. With this study we are looking to introduce a better and safer way to exercise for people with osteoarthritis and obesity. The results of this study will also allow for further development of home-based exercise and telemedicine.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 75 years;
* BMI ≥ 30.0 kg/m2 and ≤ 50.0 kg/m2;
* Symptomatic knee OA (defined as a self- report of physician diagnosis of knee OA and current knee symptoms in at least one knee determined from a minimum score of 5 of 20 on the pain subscale of the WOMAC).
* Sedentary (not meeting ACSM guidelines for physical activity)
* Medical clearance for participation

Exclusion Criteria:

* Self- reported fibromyalgia, rheumatoid arthritis, or other systemic rheumatic disease.
* Severe dementia or other memory loss condition
* Active diagnosis of psychosis or current uncontrolled substance abuse disorder
* Has been hospitalized for a stroke, heart attack, or heart failure, or had surgery for blocked arteries in the past 3 months
* Had a total joint replacement knee surgery, other knee surgery, meniscus tear, or anterior cruciate ligament tear in the past 6 months
* Is on a waiting list for total joint replacement
* Had an intra-articular injection in past 3 months or scheduled during the study period;
* Has severely impaired hearing or speech
* Is pregnant
* Has a serious or terminal illness as indicated by referral to hospice or palliative care
* Resides in a nursing home
* Has any other health problems that would prohibit safe participation in the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness | Pre - Post 12 weeks
  Cardiorespiratory fitness will be quantified as peak oxygen consumption (VO2max) and walking efficiency. VO2max will be evaluated using a Balke treadmill exercise testing protocol [35]. This protocol maintains a constant speed during the test and progressively increases treadmill inclination (grade) until exhaustion. In contrast, walking efficiency will be evaluated using a submaximal exercise test (performed prior to the VO2max test). This submaximal exercise test will require participants to walk on a treadmill at a self-selected pace, during which time VO2 will be recorded.
Resting Cardiovascular Function | Pre - Post 12 weeks
  Cardiovascular function will be quantified by resting blood pressure, heart rate, heart rate variability (HRV) and carotid-femoral pulse wave velocity (cfPWV). Blood pressure and heart rate will first be collected in the seated position using a manual sphygmomanometer according to the World Health Organization (WHO) recommendations. Next, heart rate will be recorded for approximately 10 minutes in the supine position, which will be used for assessment of HRV. During this collection period, participants will breathe at a rate of approximately 7 breaths per minute, which will be maintained using a metronome. The ECG data collected during this ten-minute period will then be analyzed using time domain HRV analysis and spectral HRV analysis. Lastly, cfPWV will be collected using applanation tonometry.
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Pre - Post 12 weeks
  Subscales for pain, stiffness and physical function will be used to assess knee osteoarthritis symptomatic burden. The WOMAC includes a total of 24 items with subscales of pain (five items), stiffness (two items), and function (17 items), which are all rated on a Likert scale of 0 (no symptoms) to 4 (extreme symptoms). The total WOMAC score will be calculated (score range of 0- 96 [no to extreme problems]), as well as the pain (score 0- 20), stiffness (score 0- 8), and function (score 0- 68) subscales.
Physical function | Pre - Post 12 weeks
  The 6-minute walk test (6MWT)
Balance | Pre - Post 12 weeks
  Single leg stance time (the ability to stand on one limb unassisted) will be recorded in seconds (maximum time = 30 seconds) [43]. Three trials will be completed using an AMTI force platform (AMTI OPT464508HF sampling at 1000Hz; AMTI, USA) to assess postural balance control in quiet bipedal stance. Participants will stand as still as possible in a relaxed upright position with their feet parallel on predetermined marks (10 cm apart) and with their arms hanging against the thighs. Center of pressure displacement will be measured under two conditions: 1) eyes open; and 2) eyes closed. In the eyes open condition, participants will be asked to look at a target 2.5 m in front of them. In the eyes closed condition, a blindfold will be used to assure the absence of visual feedback.
Muscle Strength | Pre - Post 12 weeks
  A Biodex isokinetic dynamometer (Biodex, Corp., Shirley, NY) will be used to measure the isometric strength of knee flexors and extensors.
Body Composition | Pre - Post 12 weeks
  Whole-body and appendicular body (i.e., arms and legs) composition parameters including total fat mass, fat-free mass, body fat percent, and bioelectrical impedance (lower-body segmental extracellular and intracellular water content, resistance, reactance) will be performed throughout the intervention to assess tissue level improvements in body composition components specific to the desired outcomes of the intervention.
Fasting Blood Glucose | Pre - Post 12 weeks
  FBG will be collected at baseline prior to the intervention and again at weeks 6 and 12. For measurements of FBG, participants will arrive at the laboratory after an overnight fast from food (≥ 8 hours) and abstention from exercise (≥ 12 hour). Upon arrival, participants FBG will be collected from capillary blood using a standard glucometer (KetoMojo, Napa, California, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- University Southern Mississippi, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Undecided